CLINICAL TRIAL: NCT00740220
Title: Reproducibility of 6 Minute Walk Tests for Oxygen Desaturation
Acronym: 6MWT
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: BG02-489
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Results first posted 2009-04-20 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2016-04

CONDITIONS: Hypoxemia; Anoxia; Chronic Obstructive Pulmonary Disease
Keywords: hypoxemia; anoxia; oxygen; dyspnea; pulmonary disease; chronic obstructive
MeSH Terms: conditions — Hypoxia; Pulmonary Disease, Chronic Obstructive; Dyspnea; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Each subject will be their own control. Each subject will perform three 6MWTs. Intra-subject reproducibility is being tested.

SUMMARY:
This trial will test the hypothesis that the 6 minute walk test (6MWT) is not reproducible as a measure for oxygen desaturation.

DETAILED DESCRIPTION:
Over 16 million adults in the United States are afflicted with chronic obstructive pulmonary disease (COPD) and is the fourth leading cause of death.(McCrory et al. 1190-209). COPD accounts for direct health-care costs of $18 billion.(McCrory et al. 1190-209). Oxygen therapy has been shown to decrease mortality in COPD patients with severe hypoxemia at rest. Oxygen therapy now accounts for the number one expenditure for durable medical equipment. Current requirements for oxygen therapy for COPD patients include a resting or exercise paO2 or spO2 of 55 mmHg or 88% respectively. We have shown that a resting spO2 of < 95% is predictive of those at risk of exercise induced hypoxemia in COPD patients(Knower et al. 732-36) based on continuous spO2 monitoring during a 6 minute walk. Although, the reproducibility of a 6 minute walk has been addressed in terms of a hospital test, simulated home test and actual home test (Guyatt), its inter-variability is not well studied.

We propose to investigate the reliability and inter-variability of the 6 minute walk for oxygen prescription. Currently, two programs are providing pulmonary rehabilitation for COPD patients in the community. Patients perform 6 minute walks under supervision and are monitored by pulse oximetry on a routine basis as part of these programs. We plan to capture the oximetry data in order to determine the reliability of oxygen prescriptions using the 6 minute walk. Patients who are performing a 6 minute walk will be eligible for enrollment. Protocols for the 6 minute walk are already in place and approved by their respective authority in both of the Pulmonary Rehabilitation Programs. These patients will have repeat 6 minute walks on separate in close proximity to determine the reliability of spO2 on any given day. Statistical analysis will be done by the kappa statistic for inter-test agreement in a 3 dimensional matrix.

We ask to waive consent for this study as there is no change to the daily routine of the 6 minute walks already being done as part of Pulmonary Rehabilitation. We plan only to capture the data from these walks.

ELIGIBILITY:
Inclusion Criteria:

* Taking part in Pulmonary Rehabilitation

Exclusion Criteria:

* Inability to perform 6MWT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be carried out in a population of subjects who are taking part in Pulmonary Rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2006-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arjun B Chatterjee, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data could only be shared if requestor had IRB approval and funding to re-contact all participants for permission.

REFERENCES:
- [Background] Guyatt GH, McKim DA, Weaver B, Austin PA, Bryan RE, Walter SD, Nonoyama ML, Ferreira IM, Goldstein RS. Development and testing of formal protocols for oxygen prescribing. Am J Respir Crit Care Med. 2001 Mar;163(4):942-6. doi: 10.1164/ajrccm.163.4.2002135. PMID 11282770
- [Background] Knower MT, Dunagan DP, Adair NE, Chin R Jr. Baseline oxygen saturation predicts exercise desaturation below prescription threshold in patients with chronic obstructive pulmonary disease. Arch Intern Med. 2001 Mar 12;161(5):732-6. doi: 10.1001/archinte.161.5.732. PMID 11231707
- [Background] McCrory DC, Brown C, Gelfand SE, Bach PB. Management of acute exacerbations of COPD: a summary and appraisal of published evidence. Chest. 2001 Apr;119(4):1190-209. doi: 10.1378/chest.119.4.1190. PMID 11296189
- [Background] Long term domiciliary oxygen therapy in chronic hypoxic cor pulmonale complicating chronic bronchitis and emphysema. Report of the Medical Research Council Working Party. Lancet. 1981 Mar 28;1(8222):681-6. PMID 6110912
- [Background] Continuous or nocturnal oxygen therapy in hypoxemic chronic obstructive lung disease: a clinical trial. Nocturnal Oxygen Therapy Trial Group. Ann Intern Med. 1980 Sep;93(3):391-8. doi: 10.7326/0003-4819-93-3-391. PMID 6776858
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Bradley JM, O'Neill B. Short-term ambulatory oxygen for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2005 Oct 19;2005(4):CD004356. doi: 10.1002/14651858.CD004356.pub3. PMID 16235359
- [Background] Casanova C, Cote C, Marin JM, Pinto-Plata V, de Torres JP, Aguirre-Jaime A, Vassaux C, Celli BR. Distance and oxygen desaturation during the 6-min walk test as predictors of long-term mortality in patients with COPD. Chest. 2008 Oct;134(4):746-752. doi: 10.1378/chest.08-0520. Epub 2008 Jul 14. PMID 18625667
- [Background] Celli BR, Cote CG, Marin JM, Casanova C, Montes de Oca M, Mendez RA, Pinto Plata V, Cabral HJ. The body-mass index, airflow obstruction, dyspnea, and exercise capacity index in chronic obstructive pulmonary disease. N Engl J Med. 2004 Mar 4;350(10):1005-12. doi: 10.1056/NEJMoa021322. PMID 14999112
- [Background] Croxton TL, Bailey WC. Long-term oxygen treatment in chronic obstructive pulmonary disease: recommendations for future research: an NHLBI workshop report. Am J Respir Crit Care Med. 2006 Aug 15;174(4):373-8. doi: 10.1164/rccm.200507-1161WS. Epub 2006 Apr 13. PMID 16614349
- [Background] Drummond MB, Blackford AL, Benditt JO, Make BJ, Sciurba FC, McCormack MC, Martinez FJ, Fessler HE, Fishman AP, Wise RA; NETT Investigators. Continuous oxygen use in nonhypoxemic emphysema patients identifies a high-risk subset of patients: retrospective analysis of the National Emphysema Treatment Trial. Chest. 2008 Sep;134(3):497-506. doi: 10.1378/chest.08-0117. Epub 2008 Jul 18. PMID 18641094
- [Background] Dunne PJ. The demographics and economics of long-term oxygen therapy. Respir Care. 2000 Feb;45(2):223-8; discussion 228-30. PMID 10771794
- [Background] Eaton T, Young P, Milne D, Wells AU. Six-minute walk, maximal exercise tests: reproducibility in fibrotic interstitial pneumonia. Am J Respir Crit Care Med. 2005 May 15;171(10):1150-7. doi: 10.1164/rccm.200405-578OC. Epub 2005 Jan 7. PMID 15640367
- [Background] Eiser N, Willsher D, Dore CJ. Reliability, repeatability and sensitivity to change of externally and self-paced walking tests in COPD patients. Respir Med. 2003 Apr;97(4):407-14. doi: 10.1053/rmed.2002.1462. PMID 12693802
- [Background] Emtner M, Porszasz J, Burns M, Somfay A, Casaburi R. Benefits of supplemental oxygen in exercise training in nonhypoxemic chronic obstructive pulmonary disease patients. Am J Respir Crit Care Med. 2003 Nov 1;168(9):1034-42. doi: 10.1164/rccm.200212-1525OC. Epub 2003 Jul 17. PMID 12869359
- [Background] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683
- [Background] Escourrou PJ, Delaperche MF, Visseaux A. Reliability of pulse oximetry during exercise in pulmonary patients. Chest. 1990 Mar;97(3):635-8. doi: 10.1378/chest.97.3.635. PMID 2106411
- [Background] Garcia-Talavera I, Garcia CH, Macario CC, de Torres JP, Celli BR, Aguirre-Jaime A. Time to desaturation in the 6-min walking distance test predicts 24-hour oximetry in COPD patients with a PO2 between 60 and 70mmHg. Respir Med. 2008 Jul;102(7):1026-32. doi: 10.1016/j.rmed.2008.02.004. Epub 2008 Mar 17. PMID 18343649
- [Background] Guyatt GH, Nonoyama M, Lacchetti C, Goeree R, McKim D, Heels-Ansdell D, Goldstein R. A randomized trial of strategies for assessing eligibility for long-term domiciliary oxygen therapy. Am J Respir Crit Care Med. 2005 Sep 1;172(5):573-80. doi: 10.1164/rccm.200412-1692OC. Epub 2005 May 18. PMID 15901604
- [Background] Guyatt GH, McKim DA, Austin P, Bryan R, Norgren J, Weaver B, Goldstein RS. Appropriateness of domiciliary oxygen delivery. Chest. 2000 Nov;118(5):1303-8. doi: 10.1378/chest.118.5.1303. PMID 11083678
- [Background] Hadeli KO, Siegel EM, Sherrill DL, Beck KC, Enright PL. Predictors of oxygen desaturation during submaximal exercise in 8,000 patients. Chest. 2001 Jul;120(1):88-92. doi: 10.1378/chest.120.1.88. PMID 11451821
- [Background] Lewis CA, Eaton TE, Fergusson W, Whyte KF, Garrett JE, Kolbe J. Home overnight pulse oximetry in patients with COPD: more than one recording may be needed. Chest. 2003 Apr;123(4):1127-33. doi: 10.1378/chest.123.4.1127. PMID 12684303
- [Background] MacIntyre NR. Oxygen therapy and exercise response in lung disease. Respir Care. 2000 Feb;45(2):194-200; discussion 201-3. PMID 10771791
- [Background] Mak VH, Bugler JR, Roberts CM, Spiro SG. Effect of arterial oxygen desaturation on six minute walk distance, perceived effort, and perceived breathlessness in patients with airflow limitation. Thorax. 1993 Jan;48(1):33-8. doi: 10.1136/thx.48.1.33. PMID 8434350
- [Background] McGovern JP, Sasse SA, Stansbury DW, Causing LA, Light RW. Comparison of oxygen saturation by pulse oximetry and co-oximetry during exercise testing in patients with COPD. Chest. 1996 May;109(5):1151-5. doi: 10.1378/chest.109.5.1151. PMID 8625659
- [Background] O'Donohue WJ Jr, Plummer AL. Magnitude of usage and cost of home oxygen therapy in the United States. Chest. 1995 Feb;107(2):301-2. doi: 10.1378/chest.107.2.301. No abstract available. PMID 7842750
- [Background] Poulain M, Durand F, Palomba B, Ceugniet F, Desplan J, Varray A, Prefaut C. 6-minute walk testing is more sensitive than maximal incremental cycle testing for detecting oxygen desaturation in patients with COPD. Chest. 2003 May;123(5):1401-7. doi: 10.1378/chest.123.5.1401. PMID 12740254
- [Background] Romagnoli M, Dell'Orso D, Lorenzi C, Crisafulli E, Costi S, Lugli D, Clini EM. Repeated pulmonary rehabilitation in severe and disabled COPD patients. Respiration. 2006;73(6):769-76. doi: 10.1159/000092953. Epub 2006 Apr 21. PMID 16636528
- [Background] Rooyackers JM, Dekhuijzen PN, Van Herwaarden CL, Folgering HT. Training with supplemental oxygen in patients with COPD and hypoxaemia at peak exercise. Eur Respir J. 1997 Jun;10(6):1278-84. doi: 10.1183/09031936.97.10061278. PMID 9192929
- [Background] Sciurba F, Criner GJ, Lee SM, Mohsenifar Z, Shade D, Slivka W, Wise RA; National Emphysema Treatment Trial Research Group. Six-minute walk distance in chronic obstructive pulmonary disease: reproducibility and effect of walking course layout and length. Am J Respir Crit Care Med. 2003 Jun 1;167(11):1522-7. doi: 10.1164/rccm.200203-166OC. Epub 2003 Feb 20. PMID 12615634
- [Background] Timms RM, Kvale PA, Anthonisen NR, Boylen CT, Cugell DW, Petty TL, Williams GW. Selection of patients with chronic obstructive pulmonary disease for long-term oxygen therapy. JAMA. 1981 Jun 26;245(24):2514-5. PMID 7014957
- [Background] Ram FS, Wedzicha JA. Ambulatory oxygen for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2002;(2):CD000238. doi: 10.1002/14651858.CD000238. PMID 12076387
- [Background] Zielinski J, Tobiasz M, Hawrylkiewicz I, Sliwinski P, Palasiewicz G. Effects of long-term oxygen therapy on pulmonary hemodynamics in COPD patients: a 6-year prospective study. Chest. 1998 Jan;113(1):65-70. doi: 10.1378/chest.113.1.65. PMID 9440570
- [Background] Budweiser S, Heidtkamp F, Jorres RA, Heinemann F, Arzt M, Schroll S, Schmidbauer K, Hitzl AP, Pfeifer M. Predictive significance of the six-minute walk distance for long-term survival in chronic hypercapnic respiratory failure. Respiration. 2008;75(4):418-26. doi: 10.1159/000109662. Epub 2007 Oct 9. PMID 17934248

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Prospective Observational Study: Each subject will be their own control. Each subject will perform three 6MWTs. Intra-subject reproducibility is being tested. These will all be subjects in Pulmonary Rehab.
Period: Overall Study
Arm/Group | Single Arm Prospective Observational Study
Started | 97
Completed | 88
Not Completed | 9
Not completed — screen failures (non-COPD patients) | 9

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Prospective Observational Study
Number analyzed (Participants) | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 97

OUTCOME MEASURES:

1. Primary Outcome: Kappa Statistic for Correlation of the Oxygen Saturation Across 3 Serial 6 Minute Walk Tests (6MWT)
Description: The kappa statistic is a measure of the quality of a test. It is a ratio.
Time Frame: All three 6MWTs should take place within 30 days
Measure: Number; unit: Ratio
Arm/Group | Single Arm Prospective Observational Study
Number analyzed (Participants) | 88
Ratio | 0.62

ADVERSE EVENTS:
Arm/Group | Single Arm Prospective Observational Study
Serious Adverse Events (participants affected / at risk) | 0/88
Other Adverse Events (participants affected / at risk) | 0/88

LIMITATIONS AND CAVEATS:
Study was conducted in a Pulmonary Rehabilitation Population and may not be generalizable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No